CLINICAL TRIAL: NCT00375271
Title: Multicenter Randomized Controled Trial of Perioperative Hemodynamic Optimization in High-Risk Patients Using Less-Invasive Monitoringng Methods
Brief Title: Perioperative Hemodynamic Optimization in High-Risk Patients Using Less-Invasive Monitoring Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro de Estudos Mário César de Rezende (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONEP 12523; 25000.185884/2005-15
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2006-09

CONDITIONS: Postoperative Care
Keywords: Monitoring, Intraoperative; Hemodynamic Processes; Treatment Protocols

INTERVENTIONS:
Procedure: perioperative hemodynamic optimization protocol

SUMMARY:
The aim of this study is to evaluate different strategies of hemodynamic optimization in high risk surgical patients during the first twelve postoperative hours in ICU based on a protocol guided by a less invasive monitorig tool (Vigileo®), oriented by a fiberoptic central venous catheter that allows continuous monitorig of SvcO2 (PreSep®), and a pressure transducer (FloTrac®) that allows cardiac output calculation by the standard deviation of mean arterial pressure or a standard resuscitation strategy.

DETAILED DESCRIPTION:
Patients submitted to high risk surgical procedures generally show a hyperdynamic pattern due to the metabolic response after the surgical trauma. This response is fundamentally dependent on their functional reserve and on the treatment. Data from UK show an aged population with 15 to 30% of mortality in the first thirty days after surgery, generally having respiratory or cardiac co-morbidities1. Identification of these patients besides protocol implementation aiming to an appropriate support is the basic strategy to warrant a better outcome in the post-operative period.

Shoemaker has established the definition criteria to high risk patients at the end of the 80's. Those criteria are accepted until today. He too demonstrated the benefits of hemodynamic optimization in order to achieve "supra-normal" oxygen delivery.

Unfortunately, in the years to come, there was a backlash in this concept due to results of several heterogeneous and misleading studies that cast doubts about the efficacy of that strategy. Heyland, however, observed benefit when the hemodynamic optimization was instituted before the surgery.

In the 90's, support to high risk surgical patients had a new start, with publication of several studies demonstrating reduction on morbidity, mortality, and hospital and ICU lengths of stay. In a recent metaanalysis of twenty one studies, Kern and Shoemaker concluded that there was mortality reduction when hemodynamic optimization was started early before organ dysfunction has ensued. There was greater benefit in those studies where the control group had a 20% mortality or more and when the therapy achieved differences on oxygen delivery between the control and treatment groups.

Despite the strong evidence favoring hemodynamic optimization, as long as the high risk patients are identified, more studies are necessary to better answer some questions such as: what is the importance of volemic replacement, what is the best solution to be used, and what is the best method for monitoring for the patient response. Catecholamines must be used carefully, despite their theoretic capacity of modulating inflammatory response. It appears that optimization has to be done early in the pre-operative period when organ dysfunction has not ensued yet. We have to discover for how long the optimization has to be maintained during and after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* High risk elective surgeries* according to adapted Shoemaker criteria.
* Request of post-operative support by the surgeon and anesthetist.
* Patients that have need of central venous and arterial catheters according to surgeon, critical care physician or anesthetist evaluation.
* Informed consent will be obtained from all patients enrolled or their next of kin.

Exclusion Criteria:

* Patients with terminal disease, submitted to palliative surgery;
* Cardiac failure class IV of NYHA;
* Chronic renal failure without dyalisis and intolerant to fluids;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2006-08; Study Completion 2007-06

PRIMARY OUTCOMES:
60 days mortality

SECONDARY OUTCOMES:
Organ dysfunction by means of SOFA score,
Postoperative complications, and
ICU and hospital lenghts of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Ederlon Rezende, MD, Study Chair — Hospital do Servidor Publico Estadual; Álvaro Réa-Neto, MD, Principal Investigator — Hospital de Clínicas da Universidade Federal do Paraná; Ciro L Mendes, MD, Principal Investigator — Hospital Universitário da Universidade Federal da Paraíba; Fernando S Dias, MD, Principal Investigator — Hospital São Lucas da Pontifice Universidade Católica do Rio Grande do Sul; José Eduardo C Castro, MD, Principal Investigator — Hospital Copa D'Or; Rubens C Costa Filho, MD, Principal Investigator — Hospital Procardíaco; Suzana Margareth A Lobo, MD, Principal Investigator — Hospital de Base da Faculdade de Medicina de São José do Rio Preto
Locations (1):
- Hospital do Servidor Público Estadual, São Paulo, São Paulo, Brazil